CLINICAL TRIAL: NCT05594069
Title: Effect of Triple Pre-rehabilitation on Radiotherapy for Head and Neck Cancer Patients: a Randomized Controlled Trial
Brief Title: Effect of Triple Pre-rehabilitation on Radiotherapy for Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: China International Medical Foundation (Other)
Responsible Party: Principal Investigator, luqian@bjmu.edu.cn, professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pre-rehabilitation
Record Dates: First submitted 2022-10-14; First posted 2022-10-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Triple Pre-rehabilitation; Radiotherapy; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre Group (Experimental): intervention before and during radiotherapy
  Interventions: Other: triple pre-rehabilitation; Other: triple rehabilitation
- Re Group (Other): intervention during radiotherapy only
  Interventions: Other: triple rehabilitation

INTERVENTIONS:
Other: triple pre-rehabilitation — The triple intervention consisted of exercise, nutrition and psychology. Based on the intervention framework, face-to-face intervention adjustment and intensive intervention measures were carried out from the time of enrollment (T0). Combined with weekly telephone follow-up during the intervention, the intervention content formulated face-to-face last time was reviewed, reinforcement behaviors were performed, and questions were answered during the intervention.
  Arms: Pre Group
Other: triple rehabilitation — The triple intervention consisted of exercise, nutrition and psychology. Based on the intervention framework, face-to-face intervention adjustment and intensive intervention measures were carried out at the time of the beginning of radiotherapy (T1), and the middle stage of radiotherapy (T2). Combined with weekly telephone follow-up during the intervention, the intervention content formulated face-to-face last time was reviewed, reinforcement behaviors were performed, and questions were answered during the intervention.

SUMMARY:
To evaluate the intervention effect of triple pre-rehabilitation on head and neck cancer patients with radiotherapy, and process evaluation to further optimize the intervention program.

The pre-rehabilitation intervention was develped previously based on the process of evidence-based-nursing, including interventions of nurtrtion, exercise, and psychology.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ age < 75 years old
* The pathological diagnosis of HNC included nasopharyngeal cancer, oral cancer, oropharyngeal cancer, hypopharyngeal cancer, laryngeal cancer, salivary gland cancer;
* Plan to receive radiotherapy
* Basic communication skills
* Volunteer to participate in this study.

Exclusion Criteria:

* Combined with other malignant tumors
* Distant metastasis
* Inability to measure body composition, such as metal in the body or inability to stand alone
* With contraindications to exercise (such as cardiovascular and cerebrovascular diseases, respiratory diseases, etc)
* Complicated with severe liver and kidney function damage
* Previous diagnosis of other cancers
* pregnant or lactation women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Critical weight loss | About 6 weeks
  Weight loss over 5% during radiotherapy

SECONDARY OUTCOMES:
Rate of adverse reactions of radiotherapy assessed by CTCAE v5.0 | About 6 weeks
  Adverse reactions of radiotherapy
Physical performance | About 6 weeks
  Physical performance measured by the 4-Meter Walk Test
Physical performance | About 6 weeks
  Physical performance measured by 30-Second Chair Stand Test (30-SCST)
Physical performance | About 6 weeks
  Physical performance measured by hand grip strength
Body composition measured by Bioelectrical Impedance Analysis (BIA) | About 6 weeks
  Body composition measured by Bioelectrical Impedance Analysis (BIA)
Quality of life of patients assessed by QLQ-C30 | About 6 weeks
  Quality of life of patients assessed by QLQ-C30
Intake assessed by a simple diet self-assessment tool (SDSAT) | About 6 weeks
  Intake assessed by a simple diet self-assessment tool (SDSAT)
Psychological status assessed by hospital anxiety and depression scale (HADS) | About 6 weeks
  Psychological status assessed by hospital anxiety and depression scale (HADS)
Number of participants with intervention-related adverse events | About 6 weeks
  Number of participants with intervention-related adverse events
Patients in the intervention group were interviewed about the compliance of the study | About 6 weeks
  Patients in the intervention group were interviewed about the compliance of the study
Patients in the intervention group were interviewed about the experience of the study | About 6 weeks
  Patients in the intervention group were interviewed about the experience of the study

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, Professor, Study Chair — School of Nursing Peking University
Locations (1):
- Tianjin medical university cancer institute and hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT05594069/ICF_000.pdf